CLINICAL TRIAL: NCT06188026
Title: Investigation of the Effect of NNC0194-0499 on Pharmacokinetics of a Combined Oral Contraceptive (Ethinylestradiol and Levonorgestrel) in Females of Non-childbearing Potential. .
Brief Title: A Research Study Looking at How the Compound NNC0194-0499 Works With Birth Control Pills in Women Not Able to Bear Children.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NN9500-4619; U1111-1279-3843 (Other: World Health Organization (WHO)); 2023-503595-24-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-12-14; First posted 2024-01-03 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteers (Non-alcoholic Steatohepatitis)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Ethinyl Estradiol; Levonorgestrel

STUDY DESIGN:
Intervention Model Description: single-centre, one-sequence cross-over, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequence 1 (Experimental): All participants will be exposed to both interventions in a defined sequence. OC 8 days, NNC0194-0499 4 weeks, OC/NNC0194-0499 combined 1 week.
  Interventions: Drug: NNC0194-0499; Drug: ethinylestradiol/levonorgestrel

INTERVENTIONS:
Drug: NNC0194-0499 — Once a week for 5 weeks as an injection in dose of 30 mg. The injection will be given under the skin
Drug: ethinylestradiol/levonorgestrel — Oral contraceptive is taken as tablet daily composed of 30 μg ethinylestradiol and 150 μg levonorgestrel.

SUMMARY:
The study will investigate the influence of NNC0194-0499 on the blood levels of the two components of a birth control pill, Microgynon®. Participants will get the birth control pill in form of tablets in two periods of 8 days each.

Participants will get NNC0194-0499 as injection under the skin of their thigh. The injections will be given once weekly for 5 weeks.

The study will last for about 11 to 15 weeks, depending on the length of the screening period.

Participants will have to stay overnight at the study centre (2 nights and 4 nights, respectively) Only healthy women who are not able to bear children can take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* Female of non-childbearing potential.
* Age 18-65 years (both inclusive) at the time of signing the informed consent.
* Body mass index (BMI) between 18.5 and 29.9 kg/m^2 (both inclusive) at screening.
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Any disorder which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Any contraindications for the use of the oral contraception used in the study according to the Prescription Drug Information.
* Sitting blood pressure at screening outside the range of 90-139 mmHg for systolic or 50-89 mmHg for diastolic.
* Pulse outside the range of 50-89 beats/minute at screening
* Use of prescription medicinal products or non-prescription drugs including any herbal medicine known to interfere with the metabolic CYP pathways, such as hypericum (St. John's Wort), ginseng, garlic, milk thistle, and echinaceae, within 14 days before screening. Exceptions are: use of routine vitamins (vitamins used within a normal dose reference interval), occasional use of paracetamol, non-steroidal anti-inflammatory drugs (NSAIDs), or topical medication not reaching systemic circulation.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, gastrointestinal, or endocrinological conditions.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
(AUC0-24h,EE,SS), area under the ethinylestradiol plasma concentration-time curve during a dosing interval at steady state | Day 8 (pre-dose to 24 hours post-dose) and Day 38 (pre-dose to 24 hours post-dose)
  h-pg/mL
(AUC0-24h,LN,SS), area under the levonorgestrel plasma concentration-time curve during a dosing interval at steady state | Day 8 (pre-dose to 24 hours post-dose) and Day 38 (pre-dose to 24 hours post-dose)
  h-pg/mL

SECONDARY OUTCOMES:
(Cmax,EE,SS), maximum concentration of ethinylestradiol at steady state | Day 8 (pre-dose to 24 hours post-dose) and Day 38 (pre-dose to 24 hours post-dose)
  pg/mL
(Cmax,LN,SS), maximum concentration of levonorgestrel at steady state | Day 8 (pre-dose to 24 hours post-dose) and Day 38 (pre-dose to 24 hours post-dose)
  pg/mL
(tmax,EE,SS), time to maximum concentration of ethinylestradiol at steady state | Day 8 (pre-dose to 24 hours post-dose) and Day 38 (pre-dose to 24 hours post-dose)
  hours
(tmax,LN,SS), time to maximum concentration of levonorgestrel at steady state | Day 8 (pre-dose to 24 hours post-dose) and Day 38 (pre-dose to 24 hours post-dose)
  hours
Number of treatment emergent adverse events (TEAEs) | Day 1 to Day 8, and Day 31 to Day 38.
  Number of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com